CLINICAL TRIAL: NCT04585126
Title: Effect of Ultrasound-guided Intermediate Cervical Block on Recurrent Laryngeal Nerve Monitoring During Thyroid Surgery : a Randomised Non-inferiority Study
Brief Title: Effect of Cervical Block on Recurrent Laryngeal Nerve Monitoring During Thyroid Surgery
Acronym: THYRODOUL2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Collaborators: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 19-105
Record Dates: First submitted 2020-10-02; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Thyroid Surgery
Keywords: thyroid surgery; cervical nerve block; recurrent laryngeal nerve monitoring; enhanced recovery after surgery

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, double blinded, non inferiority study comparing general anesthesia combined with cervical nerve block vs general anesthesia alone in thyroid surgery
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, surgeons and outcomes assessor are blind Only the anesthesiologist taking care of the patient knows the allocation group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General anesthesia without intermediate cervical block (No Intervention): General anesthesia performed by the anesthesiologist
- General anesthesia with intermediate cervical block (Active Comparator): General anesthesia performed by the anesthesiologist associated with an echoguided intermediate cervical block (bilateral in total thyroidectomy, unilateral in partial thyroidectomy) : 10 to 30cc of ropivacaine (2 to 3,75 %)
  Interventions: Drug: Intermediate cervical block

INTERVENTIONS:
Drug: Intermediate cervical block — Local anesthesia performed in addition to the general anesthesia
  Arms: General anesthesia with intermediate cervical block

SUMMARY:
Non-inferiority study aimed to assess the impact of cervical block on recurrent laryngeal nerve monitoring during thyroid surgery Secondary outcomes will assess post-operative recovery, post-operative pain and post-operative dysphonia

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18, able to give consent after clear and fair information
* Affiliated to social security
* Total thyroidectomy performed in the context of Graves' disease in biological euthyroidism with the need for surgical treatment (pregnancy project, fluctuating TSH, etc.), or multiheteronodular goiter with suspect or compressive nodules, or lobo-isthmectomy
* No previous homolateral cervical surgery
* Professional activity
* Telephone line (at home or cellular)

Exclusion Criteria:

* Patients over 18 under legal protection
* Allergy to local anesthetics
* Existence of preoperative laryngeal dysphonia or paralysis
* Patient with a submerging goiter (lower edge of the thyroid not seen on the preoperative cervical ultrasound)
* Presence of uncontrolled infectious pathology
* Pregnant or breastfeeding woman or no contraception
* Lymph node dissection planned or patient at high risk of lymph node dissection (BETHESDA 5 and 6)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Effect on recurrent laryngeal nerve monitoring | Before surgical dissection
  Percentage of bilateral and unilateral non-response to recurrent laryngeal nerve monitoring

SECONDARY OUTCOMES:
Postoperative recovery | 7 days post surgery
  Ability to return to work assessed by a composite questionnaire (QOR15 / FRI / patient's personal opinion)
Postoperative pain | First 24 hours post surgery
  Numerical rating pain scale (0 = no pain to 10 = worst pain)
Early postoperative complications | First 24 hours post surgery
  Number of patients with hypocalcemia, hematoma, nausea, vomiting
Postoperative dysphonia | During the first 24 hours and 7 days post surgery
  Number of patients with post-operative dysphonia
Late postoperative complications | 1 to 3 months post surgery
  Number of patients with persistent laryngeal nerve paralysis and/or dysphonia, persistent hypocalcemia, rehospitalization, revision surgery

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Babin, Principal Investigator — University Hospital, Caen
Locations (1):
- Caen University Hospital, Caen, France